CLINICAL TRIAL: NCT02890238
Title: Effect of Sildenafil Citrate on Pregnancy Rate in Women Undergoing Induction of Ovulation
Brief Title: Sildenafil Effect After Ovulation Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 156
Record Dates: First submitted 2016-08-29; First posted 2016-09-07 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Infertility
Keywords: Sildenafil Citrate; Induction of Ovulation; Pregnancy Rate
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil citrate (Active Comparator): 50 women who will be given clomiphene citrate 50mg (clomid,) orally 2times/day from 2rd - 7th day of the cycle and sildenafil citrate 20mg tab from 7th-11th day of the same cycle orally 3times/day
  Interventions: Drug: Clomiphene citrate; Drug: sildenafil citrate
- placebo group (Placebo Comparator): 50 women who will be given clomiphene citrate 50mg (clomid,) orally 2times/day from 2rd- 7th day of the cycle and placebo tablets from 7th-11th day of the same cycle orally 3 times/day
  Interventions: Drug: Clomiphene citrate; Drug: Placebo

INTERVENTIONS:
Drug: Clomiphene citrate — 50mg (clomid,) orally 2 times/day from 2nd- 7th day of the cycle
  Other Names: clomid
Drug: sildenafil citrate — 20mg tab from 7th-11th day of the same cycle orally 3times/day
  Other Names: Viagra
  Arms: sildenafil citrate
Drug: Placebo — tab from 7th-11th day of the same cycle orally 3times/day
  Arms: placebo group

SUMMARY:
100 women with infertility classified into 2 groups.

Group A: Included 50 women who will be given clomiphene citrate 50mg (clomid) orally 2 times/day from 2rd-7th day of the cycle and sildeaynafil citrate 20mg tab from 7th-11th day of the same cycle orally 3 times/day.

Group B: Included 50 women who will be given clomiphene citrate 50mg (clomid) orally 2 times/day from 2rd-7th day of the cycle and placebo tablets from 7th-11th day of the same cycle orally 3 times/day.

DETAILED DESCRIPTION:
100 women with infertility classified into 2 groups.

Group A: Included 50 women who will be given clomiphene citrate 50mg (clomid) orally 2 times/day from 2rd-7th day of the cycle and sildeaynafil citrate 20mg tab from 7th-11th day of the same cycle orally 3 times/day.

Group B: Included 50 women who will be given clomiphene citrate 50mg (clomid) orally 2 times/day from 2rd-7th day of the cycle and placebo tablets from 7th-11th day of the same cycle orally 3 times/day.

Folliculometry was assessed by:

* Transvaginal ultrasound: It was done on day 11th of the cycle to detect number of follicles and endometrial thickness.

When the follicles reach ≥18 ml, injection of 5000 IU of HCG IM to trigger ovulation to both groups.

Pregnancy was assessed by:

* Beta HCG test: (Radioimmunoassay)

ELIGIBILITY:
Inclusion Criteria:

1. Infertile women whether it's primary or secondary infertility
2. Woman's age: (18-35 years old)
3. Menstrual cycle from (24-35 days)
4. Normal semen analysis

Exclusion Criteria:

1. Age more than 35 years old
2. Ovarian cysts
3. Abnormal hormonal profile (e.g hyperprolactinaemia)
4. Significant cardiovascular disease
5. Serious liver disease or renal failure
6. Poorly controlled diabetes mellitus

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate per cycle | 14 days after HCG triggering of ovulation
  Serum pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes